CLINICAL TRIAL: NCT07117968
Title: Evaluating the Benefit of Integrating Connected Care to Reshape the Cochlear Implant Care Pathway: a Multicenter Randomized Non-inferiority Study
Brief Title: Benefit of Connected Care for Cochlear Implant Management
Acronym: Connect IC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL24_0756
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Investigator will conduct a randomized, comparative, multicenter study. Two prospective follow-up groups of CI patients will be set up for comparison, and each patient will be followed until their 12-month post-implantation check-up. Patients in the control group will benefit from the current follow-up, as performed in their center, and those in the experimental group will integrate the new care pathway.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): Cochlear implant patients will benefit from the current first year of post-CI follow-up care provided at their own center.
  Interventions: Other: Standard-of-care
- intervention group (Experimental): Cochlear implant patients will be integrated into the new care pathway. They will be offered early activation of the implant and hybrid follow-up, including remote or in-center monitoring visits, adjustable according to the evolution of their hearing performance and comfort.
  Interventions: Other: Experimental hybrid care pathway

INTERVENTIONS:
Other: Standard-of-care — Management of the first year post-CI follow-up according to current center practices
  Arms: control group
Other: Experimental hybrid care pathway — First year post-CI follow-up including early activation of the implant and hybrid follow-up, including remote or in-center monitoring visits, adjustable according to the evolution of their hearing performance and comfort. In this new care pathway, compared with the Standard-of-care, the 2-week visit and the 9-month visit are omitted, due to early activation and remote follow-up. Visits at 1 and 6 months are the same as those in the conventional, on-site routine. Visits at 3 and 12 months will be carried out remotely by default via the remote monitoring application.
  Arms: intervention group

SUMMARY:
Some 30 hospitals in France are accredited to manage cochlear implant (CI) activity, which represents around 1,800 new patients implanted per year and an estimated active file of over 20,000 patients.

The current patient pathway meets the requirements described in 2009 for this activity. Today, however, it is inflexible, not scalable, and presents major constraints for both patients and the healthcare professionals in charge of them. In the first year post-implantation, a patient visits his or her center on average 9 times for routine follow-up. The growing demand for patients to be implanted and the need to continue monitoring patients who have already been implanted are putting a strain on the centers responsible for this activity, leading to a deterioration in the management of this condition. We need to propose a new care pathway that meets current needs, improves patient service and optimizes the workload of our teams in order to manage their entire implant cohort.

This project focuses on two areas in order to optimize the implant patient's care pathway. The first is to integrate telemonitoring into the follow-up process. Telemonitoring has already proved its worth in many therapeutic fields, and could clearly meet the needs of all those involved: Reduced time constraints, optimized on-site visits, flexibility in management, fewer people lost to follow-up... The second axis consists in optimizing the implant system activation stage, a cumbersome and complex step, by favoring early activation based on objective patient data collected intraoperatively. Reducing the variability of activation leads to earlier stabilization of settings, without compromising hearing performance.

These two approaches are currently used in some centers, but not in combination, and have been adopted routinely in some countries. The expected benefits are therefore well known, but this project has a key role to play in demonstrating the feasibility and medico-economic benefits of our French model.

This project will therefore jointly optimize early activation, made possible by objective intraoperative measurements, and patient management by integrating telemonitoring into the adult CI pathway to improve efficiency.

The aim of this project is to evaluate, in the first year of post-CI follow-up, the benefits of this new, adapted care pathway, both in terms of the organization of care and the patient's quality of life and performance.

The main hypothesis is that a new care pathway that integrates early activation and remote monitoring will enable the center to provide more flexible and adapted patient follow-up to optimize management, and thus improve quality of life without any deterioration in clinical effectiveness (hearing performance). The investigators aim to demonstrate the clinical non-inferiority of performance in noise (DTT Test) assessed at 12 months in patients benefiting from the new care pathway vs. current standard follow-up, while improving their quality of life, in a multicenter randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 or over) eligible for a cochlear implant in primary implantation according to French National Authority for Health indications
* Patients suffering from severe to profound bilateral deafness with discrimination less than or equal to 50% on voice audiometry tests using the Fournier list (or equivalent).
* Patients affiliated to the public health insurance body
* Patients who benefit from a Cochlear® system with a processor compatible with Remote Care tools
* Patients using a smartphone compatible with the Nucleus Smart application.
* Patients who have given their written informed consent to the study
* French-speaking patients

Exclusion Criteria:

* Patients already implanted and candidates for implantation of the other ear (bilateralization), or previously implanted (re-implantation).
* Patients with concomitant illnesses that are incompatible with the use of remote monitoring,
* Pregnant women
* Patients suffering from unilateral deafness with incapacitating tinnitus
* Persons under legal protection (guardianship, curators).
* Subjects taking part in other interventional research with an exclusion period still in progress at the time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Hearing performance in noise | At 12 months post-activation of the CI
  Hearing performance measured in noise using the Digit Triple Test (DTT). This value corresponds to the signal-to-noise ratio, expressed in decibel Single Number Rating, required for the subject to recognize 50% of the speech signal presented (50% intelligibility threshold in silence = Speech Reception Threshold 50 in decibel Single Number Rating).

IPD SHARING:
Plan to Share IPD: No